CLINICAL TRIAL: NCT02419378
Title: Alemtuzumab in Autoimmune Inflammatory Neurodegeneration: Mechanisms of Action and Neuroprotective Potential
Acronym: ALAIN01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UKM12_0026; U1111-1156-6489 (Other: Universal Trial Number)
Record Dates: First submitted 2015-03-31; First posted 2015-04-17 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- alemtuzumab (Experimental): Administration of 2 courses of alemtuzumab at an interval of 1 year. Course 1: Intravenous infusion of 12 mg alemtuzumab per day on 5 consecutive days.
  Course 2: Intravenous infusion of 12 mg alemtuzumab per day on 3 consecutive days.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab

SUMMARY:
Alemtuzumab is the active agent of a drug called Lemtrada®. In the European Union, Lemtrada® is approved for the treatment of a particular form of multiple sclerosis (the so called relapsing remitting form). The excellent efficacy of the drug justifies its administration albeit a high risk of considerable side effects. In this context, so called secondary (occurring after the administration of Lemtrada®) autoimmune diseases are of particular importance. In these diseases the immune system acts against structures of the body itself; the reasons are still unknown. Autoimmune diseases may even occur several years after treatment with Lemtrada®. Therefore, patients who once received the drug need to undergo intensive long term health monitoring.

This study aims to elucidate which mechanisms cause to the positive and negative effects of Lemtrada®.

The study includes patients only, who suffer from multiple sclerosis and are indicated to be treated with Lemtrada®. All patients receive the drug according to the official recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF)
2. Age 18 to 55 years old (inclusive) as of the date the ICF is signed
3. Diagnosis of MS according to the McDonald criteria 2010 and cranial MRI scan demonstrating white matter lesions attributable to MS within 10 years before Screening
4. Onset of MS symptoms (as determined by a neurologist, either at present or retrospectively) within 10 years of the date the ICF is signed
5. EDSS score 0.0 to 5.0 (inclusive) at Screening
6. Patients with (highly) active RRMS disease course indicated to receive alemtuzumab according to the following conditions (at least 1 out of 3 conditions has to be fulfilled): 1. ≥2 MS relapses within 24 months, 2. clinical (≥1 relapse) or MRI (new gadolinium enhancing lesions) disease activity under therapy with other diseasemodifying therapies, 3. severe relapse with high disease activity (≥9 T2 hyperintense Lesions and ≥1 gadolinium enhancing lesion) on MRI.
7. Completion of all vaccinations required by the applicable immunization guidelines published by "ständige Impfkommission" (STIKO)
8. History of chickenpox or positive test for antibodies against varicella zoster virus (VZV)

Exclusion Criteria:

1. Participation in another clinical trial at present or within 4 weeks of study entry. There may be exceptions at the discretion of the Investigator.
2. Has any progressive form of MS
3. Hypersensitivity to the active substance, or to any of the excipients of Lemtrada®
4. Medical, psychiatric, cognitive, or other conditions that, in the Investigator's opinion, compromise the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol, or to complete the study
5. Any disability acquired from trauma or another illness that could interfere with evaluation of disability due to MS
6. Major systemic disease or other illness that would, in the opinion of the Investigator, compromise patient safety or interfere with the interpretation of study results, e.g., current peptic ulcer disease or other conditions that may predispose to hemorrhage
7. Known bleeding disorder (e.g,. dysfibrinogenemia, factor IX deficiency, hemophilia, Von Willebrand's disease, disseminated intravascular coagulation (DIC), fibrinogen deficiency, or clotting factor deficiency)
8. Significant autoimmune disease including but not limited to immune cytopenias, rheumatoid arthritis, systemic lupus erythematosus, other connective tissue disorders, vasculitis, inflammatory bowel disease, severe psoriasis
9. History of malignancy, except basal skin cell carcinoma
10. Major psychiatric disorder that is not adequately controlled by treatment
11. Epileptic seizures that are not adequately controlled by Treatment
12. Active infection, e.g., deep-tissue infection, that the Investigator considers sufficiently serious to preclude study participation
13. In the Investigator's opinion, is at high risk for infection (e.g., indwelling catheter, dysphagia with aspiration, decubitus ulcer, history of prior aspiration pneumonia or recurrent urinary tract infection)
14. Seropositivity for human immunodeficiency virus (HIV)
15. Infection with hepatitis C Virus
16. Past or present hepatitis B infection (positive hepatitis B serology)
17. Active infection with human cytomegaly virus (HCMV), Epstein-Barr virus (EBV), varicella-zoster virus (VZV)
18. Latent tuberculosis unless effective anti-tuberculosis therapy has been completed, or active tuberculosis.
19. Invasive fungal infections in history and at present
20. Cervical cytology other than PAP I or PAP II (Papanicolaou) or cervical high risk human papillomavirus (HPV) positivity
21. Any other illness or infection (latent or active) that, in the Investigator's opinion, could be exacerbated by study medication
22. Differential blood count < lower limit of normal (LLN) at Screening
23. Confirmed platelet count < the LLN of the evaluating laboratory at Screening or documented at <100,000/μL within the past year on a sample without platelet clumping
24. Presence (i.e., above the ULN) of anti-thyroid stimulating hormone receptor antibodies (anti-TSHR) and anti-thyroid peroxidase antibody (anti-TPO)
25. Any hepatic or renal function value grade 2 or higher at Screening, with the exception of hyperbilirubinemia due to Gilbert's syndrome. See Table below, drawn from the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v4.0 (CTCAE), published 28 May 2009.

    Hepatic

    Bilirubin >1.5 × ULN

    SGOT/AST >3.0 × ULN

    SGPT/ALT >3.0 × ULN

    Alkaline phosphatase >2.5 × ULN

    Renal

    Creatinine > 1.5 × ULN
26. Vaccination less than 6 weeks prior to treatment with Lemtrada.
27. Treatment with antineoplastic or immunosuppressive drugs within 8 weeks prior to study inclusion
28. Intolerance of pulsed corticosteroids, especially a history of steroid psychosis
29. Inability to undergo MRI with gadolinium administration
30. Of childbearing potential with a positive serum pregnancy test, pregnant or lactating
31. Female patients of childbearing potential: Unwilling to agree to use a reliable and acceptable contraceptive method (Pearl index <1) throughout the study period. These methods include: hormone releasing intrauterine device (IUD), hormonal-based contraception, surgical sterilization, abstinence, or double-barrier contraception (condom and occlusive cap [diaphragm or cervical cap combined with spermicide]).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in naïve CD4 positive T cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in naïve CD4 positive T cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in naïve CD8 positive T cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in naïve CD8 positive T cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
  12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD4 positive T effector cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in CD4 positive T effector cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD8 positive T effector cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD4 positive T memory cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in CD4 positive T memory cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD8 positive T memory cell counts peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in CD8 positive T memory cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD4 positive regulatory T cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in CD4 positive regulatory T cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD8 positive regulatory T cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in CD8 positive regulatory T cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in Th1 T-helper cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in Th1 T-helper cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in Th2 T-helper cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in Th2 T-helper cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in Th17 T-helper cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in Th17 T-helper cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in recent bone marrow emigrant B cell counts peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in recent bone marrow emigrant B cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in mature naïve B cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in mature naïve B cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in memory B cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in memory B cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in plasma cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in plasma cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD56bright natural killer cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in CD56bright natural killer cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD56dim natural killer cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in CD56dim natural killer cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in natural killer T cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in natural killer T cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD303+ plasmacytoid dendritic cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in CD303+ plasmacytoid dendritic cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD11c+ myeloid dendritic cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in CD11c+ myeloid dendritic cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in CD141+ myeloid dendritic cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in CD141+ myeloid dendritic cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in monocyte counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in monocyte counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in macrophage counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in macrophage counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute change from baseline in myeloid-derived suppressor cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative change from baseline in myeloid-derived suppressor cell counts in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.

SECONDARY OUTCOMES:
Absolute change from baseline in naïve CD4 positive T cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in naïve CD4 positive T cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in naïve CD8 positive T cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in naïve CD8 positive T cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD4 positive T effector cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD4 positive T effector cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD8 positive T effector cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD8 positive T effector cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD4 positive T memory cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD4 positive T memory cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD8 positive T memory cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD8 positive T memory cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD4 positive regulatory T cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD4 positive regulatory T cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD8 positive regulatory T cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD8 positive regulatory T cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in Th1 T-helper cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in Th1 T-helper cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in Th2 T-helper cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in Th2 T-helper cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in Th17 T-helper cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in Th17 T-helper cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in recent bone marrow emigrant B cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in recent bone marrow emigrant B cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in mature naïve B cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in mature naïve B cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in memory B cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in memory B cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in plasma cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in plasma cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD56bright natural killer cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD56bright natural killer cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD56dim natural killer cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD56dim natural killer cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in natural killer T cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in natural killer T cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD303+ plasmacytoid dendritic cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD303+ plasmacytoid dendritic cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD11c+ myeloid dendritic cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD11c+ myeloid dendritic cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in CD141+ myeloid dendritic cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in CD141+ myeloid dendritic cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in monocyte counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in monocyte counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in macrophage counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in macrophage counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Absolute change from baseline in myeloid-derived suppressor cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative change from baseline in myeloid-derived suppressor cell counts in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Activation status of cell surface receptors on T cells fom peripheral blood as assessed by flow cytometry | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
  Relative and absolute change from baseline of mean fluorescence intensity (MFI) and of proportion of positive cells regarding CD25, HLA-DR, LFA-1, CD29, CD69, CD71 expression
Activation status of cell surface receptors on T cells from cerebrospinal fluid as assessed by flow cytometry | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
  Relative and absolute change from baseline of mean fluorescence intensity (MFI) and of proportion of positive cells regarding CD25, HLA-DR, LFA-1, CD29, CD69, CD71 expression
Expression of co-inhibitory molecules by T cells from peripheral blood as assessed by flow cytometry | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
  Relative and absolute change from baseline of MFI and of proportion of positive cells regarding PD-1 = CD279, ICOS = CD278, TIM-3, CTLA4 expression
Expression of co-inhibitory molecules by T cells from cerebrospinal fluid as assessed by flow cytometry | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
  Relative and absolute change from baseline of MFI and of proportion of positive cells regarding PD-1 = CD279, ICOS = CD278, TIM-3, CTLA4 expression
Effector functions of CD4 and CD8 positive T cells from peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
  * Relative and absolute change from baseline of the results of cell proliferation assays assessed as percentage of proliferated cells
  * Relative and absolute change from baseline of cytokine production measurement assessed as concentration
  * Relative and absolute change from baseline of cytolytic activity assessed by flow cytometry measurement of MFI and proportion of positive cells regarding Granzyme B, Perforin and CD107a expression
  * Relative and absolute change from baseline of intracellular calcium response assessed as concentration
Effector functions of CD4 and CD8 positive T cells from cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
  * Relative and absolute change from baseline of the results of cell proliferation assays assessed as percentage of proliferated cells
  * Relative and absolute change from baseline of cytokine production measurement assessed as concentration
  * Relative and absolute change from baseline of cytolytic activity assessed by flow cytometry measurement of MFI and proportion of positive cells regarding Granzyme B, Perforin and CD107a expression
  * Relative and absolute change from baseline of intracellular calcium response assessed as concentration
Migrational capacity of T cells from peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
  * Relative and absolute change from baseline MFI and proportion of positive cells assessed by flow cytometry expression analysis of CD11a, CD31, CD44, CD49d, CCR5, CCR6, CCR7
  * Absolute and relative change of cell numbers of migrated cells compared to baseline assessed in an in vitro model by flow cytometry analysis
Migrational capacity of T cells from cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
  * Relative and absolute change from baseline MFI and proportion of positive cells assessed by flow cytometry expression analysis of CD11a, CD31, CD44, CD49d, CCR5, CCR6, CCR7
  * Absolute and relative change of cell numbers of migrated cells compared to baseline assessed in an in vitro model by flow cytometry analysis
Spectratyping of the T cell repertoire of T cells from peripheral blood concerning the expansion of distinct clones | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
  * Relative and absolute change from baseline for complexity scores
  * Qualitative comparison of the distribution of CDR3 sequences
Spectratyping of the T cell repertoire of T cells from cerebrospinal fluid concerning the expansion of distinct clones | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
  * Relative and absolute change from baseline for complexity scores
  * Qualitative comparison of the distribution of CDR3 sequences
Regulatory T-cell function in peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
  * Relative and absolute change from baseline in production of TGF-beta and IL-10 of CD4+CD25+FOXP3+ regulatory T cells
  * Suppression of T cell proliferation: Relative and absolute change from baseline in responder T cell proliferation assessed by suppression assays
Regulatory T-cell function in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
  * Relative and absolute change from baseline in production of TGF-beta and IL-10 of CD4+CD25+FOXP3+ regulatory T cells
  * Suppression of T cell proliferation: Relative and absolute change from baseline in responder T cell proliferation assessed by suppression assays
Relative and absolute change from baseline in the concentration of markers in the cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
  * S100β
  * Tau
  * phospho-Tau
  * β-Amyloid
  * Neurofilament (low weight)
  * Neurofilament (high weight)
  * N-acetylaspartate (NAA)
  * Tubulin
  * Actin
  * neuron-specific enolase (NSE)
  * glial fibrillary acidic protein (GFAP)
Relative and absolute change from baseline in neuronal activity, action potential generation and cellular integrity by obtained human CSF supernatant samples using multi-electrode arrays | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Relative and absolute change from baseline in the concentration of neurotrophic factors in the peripheral blood | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
  * Nerve growth factor (NGF)
  * brain-derived neurotrophic factor (BDNF)
  * neurotrophin-3 (NT-3)
  * and neurotrophin-4 (NT-4)
  * ciliary neurotrophic factor (CNTF)
Relative and absolute change from baseline in the concentration of neurotrophic factors in cerebrospinal fluid | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
  * Nerve growth factor (NGF)
  * brain-derived neurotrophic factor (BDNF)
  * neurotrophin-3 (NT-3)
  * and neurotrophin-4 (NT-4)
  * ciliary neurotrophic factor (CNTF)
Percent change from Baseline in the following MRI findings which are defined as markers for neurodegeneration: MRI-T1-measured cerebral volume, MRI-T1-measured number of black holes | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Relative and absolute change from baseline in retinal nerve fiber layer thickness (assessment by optical coherence tomography) | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Data on Adverse Events | Each day when the patient has a consultation with the investigator
  Clinically significant deteriorations from baseline in vital signs, results of physical examination and laboratory assessments in blood or CSF will be documented as Adverse Events

OTHER OUTCOMES:
Number of patients who experienced sustained accumulation of disability (SAD) during the study period | Date of last patient out anticipated about 4 years after study initiation
  Study period: From the day of treatment initiation until month 36 visit.
  SAD: for patients with a Baseline EDSS score of 0.0, SAD is defined as an increase of ≥1.5 points sustained over a 6-month consecutive period. For patients with a Baseline EDSS score of ≥1.0, SAD is defined as an increase of ≥1.0 point sustained over a 6-month consecutive period.
Time to SAD | At the end of each patient's study participation, i.e. 36 months after treatment initiation
Time to sustained reduction in disability (SRD) based on EDSS scores | At the end of each patient's study participation, i.e. 36 months after treatment initiation
  SRD: a ≥1 point decrease on the EDSS sustained for 6 consecutive months for patients with a baseline EDSS ≥2
Absolute Number of relapses during the study period | At the end of each patient's study participation, i.e. 36 months after treatment initiation
Number or relapses which occurred during the study period and required corticosteroid therapy | At the end of each patient's study participation, i.e. 36 months after treatment initiation
Proportion of patients who are relapse free at year 3 | Date of last patient out anticipated about 4 years after study initiation
Time to first relapse | At the end of each patient's study participation, i.e. 36 months after treatment initiation
Absolute and relative change from baseline in the following functional scores: EDSS, visual functional system score as part of the assessments for EDSS, MSFC and each MSFC component, FSMC and each subscore (mental and physical fatigue) | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 3, 6, 9, 15, 18, 21, 24, 27, 30 and 33 months after treatment initiation.
The proportion of patients who have worsened, remained stable, or improved as indicated by change from Baseline in EDSS scores at the end of the study | Date of last patient out anticipated about 4 years after study initiation
Change from baseline of the following health-related quality of life (HRQoL) measures: FAMS, EQ-5D (total score, Physical Component Summary Measure, Mental Component Summary Measure), SF-36 | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 3, 6, 9, 15, 18, 21, 24, 27, 30 and 33 months after treatment initiation.
The proportion of patients who have worsened, remained stable, or improved as indicated by change from Baseline in MSFC scores at the end of the study | Date of last patient out anticipated about 4 years after study initiation
Absolute and relative change from baseline amplitudes [V] and latencies [s] of evoked potentials (visual, somatosensory, magnetic motor evoked) | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Percent change from baseline in magnetic resonance imaging (MRI)-T2 hyperintense lesion volume | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Number of new gadolinium-enhancing lesions on MRI-T1 in comparison to Baseline | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Number of new or enlarging hyperintense lesions measured by T2-weighted MRI in comparison to Baseline | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute and relative change from baseline of IL-21 concentration in blood serum | 12, 24 and 36 months after initiation of investigational treatment. In addition on an optional basis: 6, 18 and 30 months after treatment initiation.
Absolute and relative change from baseline of following parameters assessed in CSF: cell counts, concentration of lactate, protein, and immunoglobulins (IgA, IgG, AgM) | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Qualitative assessment of the change in presence of oligoclonal bands in CSF from baseline | 12, 24 and 36 months after initiation of investigational treatment on an optional basis
Proportion of patients with no multiple sclerosis disease activity (i.e., deterioration in MRI related endpoints, relapse) at the end of the study | Date of last patient out anticipated about 4 years after study initiation

CONTACTS AND LOCATIONS:
Overall Officials: Sven Meuth, Prof. Dr. Dr., Principal Investigator — University Hospital Muenster
Locations (1):
- Universitätsklinikum Münster, Klinik für Allgemeine Neurologie, Münster, Germany

REFERENCES:
- [Derived] Ruck T, Afzali AM, Lukat KF, Eveslage M, Gross CC, Pfeuffer S, Bittner S, Klotz L, Melzer N, Wiendl H, Meuth SG. ALAIN01--Alemtuzumab in autoimmune inflammatory neurodegeneration: mechanisms of action and neuroprotective potential. BMC Neurol. 2016 Mar 10;16:34. doi: 10.1186/s12883-016-0556-9. PMID 26966029